CLINICAL TRIAL: NCT00898846
Title: Identification of the Prognostic Factors of Stage II Colon Cancer Patients Receiving Adjuvant Chemotherapy With UFT
Brief Title: Identifying Prognostic Factors in Patients Receiving Tegafur-Uracil for Stage II Colon Cancer That Was Completely Removed By Surgery
Status: Completed | Type: Observational
Sponsor: Translational Research Center for Medical Innovation, Kobe, Hyogo, Japan (Other)
Collaborators: Tokyo Medical and Dental University (Other)
Responsible Party: Sponsor
Other Study IDs: CDR0000551714; TMDU-BRI-CC-05-02
Record Dates: First submitted 2009-05-09; First posted 2009-05-12 (Estimated); Last update posted 2016-09-28 (Estimated); Status verified 2016-09

CONDITIONS: Colorectal Cancer
Keywords: stage II colon cancer; stage II rectal cancer; adenocarcinoma of the colon; adenocarcinoma of the rectum
MeSH Terms: conditions — Colorectal Neoplasms; Colonic Neoplasms; Rectal Neoplasms | interventions — Chemotherapy, Adjuvant; Tegafur

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Tumor tissue samples
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- UFT adjuvant therapy group: UFT is given at a dose of 500-600 mg/day as tegafur in 2 divided doses after meals for 5 days, followed by a 2-day rest. This one-week cycle is repeated for one year. During protocol treatment, clinical findings and laboratory values are evaluated every month. After the completion of protocol treatment, patients are followed-up, according to the schedule defined in the study protocol, for 5 years until recurrence, other malignancy or death is confirmed.
  Interventions: Drug: UFT adjuvant chemotherapy
- Observation group: Patients are followed-up without adjuvant treatment, according to the schedule defined in the study protocol, for 5 years until recurrence, other malignancy or death is confirmed.

INTERVENTIONS:
Drug: UFT adjuvant chemotherapy — UFT is given at a dose of 500-600 mg/day as tegafur in 2 divided doses after meals for 5 days, followed by a 2-day rest. This one-week cycle is repeated for one year.
  Other Names: Adjuvant chemotherapy with tegafur-uracil
  Groups: UFT adjuvant therapy group

SUMMARY:
RATIONALE: Studying samples of tumor tissue in the laboratory from patients with cancer may help doctors learn more about changes that occur in DNA and identify biomarkers related to cancer. It may also help doctors predict which patients will respond to treatment.

PURPOSE: This laboratory study is looking at prognostic factors in patients receiving tegafur-uracil for stage II colon cancer that was completely removed by surgery.

DETAILED DESCRIPTION:
OBJECTIVES:

* Identify the prognostic factors in patients with curatively resected stage II colon cancer receiving adjuvant chemotherapy with tegafur-uracil.
* Identify predictive factors of chemosensitivity to this regimen in these patients.

OUTLINE: Available tumor tissue samples are analyzed by real-time reverse transcriptase-PCR for TS, DPD, TP, OPRT, VEGF, cyclooxygenase-2, and FPGS; by PCR for microsatellite instability and genomic deletions on chromosome arm 18q; and pathologically for tumor budding, Crohn's-like lymphoid reaction, category of extent of poor differentiation, and fibrotic cancer stroma. The candidate prognostic and predictive markers are analyzed for correlation with disease-free survival, relapse-free survival, and overall survival of patients.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed adenocarcinoma of the colon or rectosigmoid

  * Stage II disease
* Must be registered on clinical trial TMDU-BRI-CC-05-01
* Must have resected tumor tissue available
* No hereditary colorectal cancer

PATIENT CHARACTERISTICS:

* ECOG performance status 0-1

PRIOR CONCURRENT THERAPY:

* Not specified

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with curatively resected stage II colon cancer in Japan.
Sampling Method: Non-Probability Sample
Enrollment: 1111 (Actual)
Dates: Start 2006-10; Primary Completion 2015-10 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
mRNA levels | 9years
  mRNA levels of patients are analyzed by the Danenberg tumor profile (DTP) method in the following indicators: thymidylate synthase (TS), dihydropyrimidine dehydrogenase (DPD), thymidine phosphorylase (TP), orotate phosphoribosyltransferase (OPRT), folylpolyglutamate synthetase (FPGS) vascular endothelial growth factor (VEGF), and cyclooxygenase-2 (Cox-2) mRNA levels.

SECONDARY OUTCOMES:
Analysis of microsatellite instability (MSI) and chromosomal instability (CIN) | At enrollment
  MSI and CIN (i.e., 18q LOH) are analyzed using paraffin embedded samples.
Histopathological examination | At enrollment
  Tumor budding, category of extent of poor differentiation, Crohn's-like lymphoid reaction, and fibrotic cancer stroma are analyzed using hematoxylin and eosin (H&E) staining of paraffin embedded samples.

CONTACTS AND LOCATIONS:
Overall Officials: Kenichi Sugihara, MD, PhD, Study Chair — Tokyo Medical and Dental University
Locations (152):
- Japan (152):
  - Nagoya Ekisaikai Hospital, Nagoya, Aichi-ken
  - Ban Buntane Houtokukai Hospital, Nagoya, Aichi-ken
  - Nagoya University Hospital, Nagoya, Aichi-ken
  - Nagoya University School of Medicine, Nagoya, Aichi-ken
  - Nagoya Midori Municipal Hospital, Nagoya, Aichi-ken
  - Aichi Prefectural Hospital, Okazaki, Aichi-ken
  - Yamamoto Kumiai General Hospital, Noshiro, Akita
  - Hiraka General Hospital, Yokote, Akita
  - Chiba Cancer Center, Chiba, Chiba
  - Teikyo University Chiba Medical Center, Ichihara, Chiba
  - Asahi General Hospital, Inba-gunn, Chiba
  - Fukuiken Saiseikai Hospital, Fukui-shi, Fukui
  - University of Fukui Hospital, Yoshida-gun, Fukui
  - National Hospital Organization Kyushu Medical Center, Fukuoka, Fukuoka
  - Kyushu University Hospital, Fukuoka, Fukuoka
  - Kitakyushu Municipal Medical Center, Kitakyushu, Fukuoka
  - Kurume University School of Medicine, Kurume, Fukuoka
  - Saint Mary's Hospital, Kurume, Fukuoka
  - Social Insurance Tagawa Hospital, Tagawa, Fukuoka
  - Fukushima Medical University Hospital, Fukushima, Fukushima
  - Gifu Municipal Hospital, Gifu, Gifu
  - Matsunami General Hospital, Gifu, Gifu
  - Hashima City Hospital, Hashima, Gifu
  - Ogaki Municipal Hospital, Ogaki-shi, Gifu
  - Gunma University Graduate School of Medicine, Maebashi, Gunma
  - Gunma Cancer Center, Otashi, Gunma
  - National Hospital Organization Fukuyama Medical Center, Fukuyama, Hiroshima
  - Chugoku Central Hospital of the Mutual Aid Association of Public School Teachers, Fukuyama, Hiroshima
  - Hiroshima University Hospital, Hiroshima, Hiroshima
  - National Hospital Organization Kure Medical Center, Kure, Hiroshima
  - Miyoshi Central Hospital, Miyoshi, Hiroshima
  - Asahikawa Medical College, Asahikawa, Hokkaido
  - Otaru Ekisaikai Hospital, Asahikawa, Hokkaido
  - Hakodate Goryoukaku Hospital, Hakodate, Hokkaido
  - Hirosaki University, School of Medicine, Otaru-shi, Hokkaido
  - Sapporo Medical University, Sapporo, Hokkaido
  - Sapporo City General Hospital, Sapporo, Hokkaido
  - Hokkaido University Graduate School of Medicine, Sapporo, Hokkaido
  - Hyogo Cancer Center, Akashi, Hyōgo
  - Ako City Hospital, Akou, Hyōgo
  - Hyogo Prefectural Amagasaki Hospital, Amagasaki, Hyōgo
  - Kansai Rosai Hospital, Amagasaki, Hyōgo
  - Himeji St. Mary's Hospital, Himeji, Hyōgo
  - Himeji Central Hospital, Himeji, Hyōgo
  - Kakogawa Municipal Hospital, Kakogawa, Hyōgo
  - Kobe University Hospital, Kobe, Hyōgo
  - Kobe City General Hospital, Kobe, Hyōgo
  - Nishi-Kobe Medical Center, Kobe, Hyōgo
  - Kobe West City Hospital, Kobe, Hyōgo
  - Kobe Medical Center, Kobe, Hyōgo
  - Sano Hospital, Kobe, Hyōgo
  - Hyogo College of Medicine, Nishinomiya, Hyōgo
  - Hyogo Prefectural Awaji Hospital, Sumoto, Hyōgo
  - Takarazuka Municipal Hospital, Takarazuka, Hyōgo
  - Higashi Takarazuka Satoh Hospital, Takarazukai, Hyōgo
  - National Hospital Organization Mito Medical Center, Ibaraki, Ibaraki
  - Kagawa University Hospital, Hiragi, Kagawa-ken
  - Kagawa Prefectural Central Hospital, Takamatsu, Kagawa-ken
  - Nanpuh Hospital, Kagoshima, Kagoshima-ken
  - Kanagawa Prefectural Ashigawa-kami Hospital, Ashigarakami-gun, Kanagawa
  - Chigasaki Municipal Hospital, Chigasaki, 253-0083, Kanagawa
  - Kitasato University School of Medicine, Kanagawa, Kanagawa
  - Kanto Rosai Hospital, Kawasaki, Kanagawa
  - Yokohama City Hospital, Yokohama, Kanagawa
  - Kanagawa Cancer Center, Yokohama, Kanagawa
  - International Goodwill Hospital, Yokohama, Kanagawa
  - Kochi Medical School, Nankoku, Kochi
  - Kumamoto University Faculty of Medical and Pharmaceutical Sciences, Kumamoto, Kumamoto
  - Japanese Red Cross Kumamoto Hospital, Kumamoto, Kumamoto
  - National Hospital Organization - Kumamotominami Hospital, Uki, Kumamoto
  - Yatsushiro Health Insurance General Hospital, Yatsushiro, Kumamoto
  - Kyoto Second Red Cross Hospital, Kanigyou-ku, Kyoto
  - Kyoto Prefectural University of Medicine, Kyoto, Kyoto
  - Nishijin Hospital, Kyoto, Kyoto
  - Mie University Graduate School of Medicine, Thu-shi, Mie-ken
  - Miyagi Cancer Center, Natori-shi, Miyagi
  - Tohoku Rosai Hospital, Sendai, Miyagi
  - Iida Municipal Hospital, Iida, Nagano
  - Showa-Inan General Hospital, Komagane, Nagano
  - Aizawa Hospital, Matsumoto, Nagano
  - Nagano Red Cross Hospital, Nagano, Nagano
  - Nagano Municipal Hospital, Nagano, Nagano
  - Hokushin Hospital, Nakano, Nagano
  - Nagasaki University Hospital, Nagasaki, Nagasaki
  - Saiseikai Nara Hospital, Nara, Nara
  - Kenseikai Nara Coloproctology Center, Yamatotakada, Nara
  - Saiseikai Niigata Daini Hospital, Niigata, Niigata
  - Niigata University Medical and Dental Hospital, Niigata, Niigata
  - Niigata Cancer Center Hospital, Niigata, Niigata
  - Oita University Hospital, Yufu-shi, Oita Prefecture
  - Kurashiki Central Hospital, Kurashiki, Okayama-ken
  - Okayama University Medical School, Okayama, Okayama-ken
  - Hoshigaoka Koseinenkin Hospital, Hirakata, Osaka
  - Rinku General Medical Center, Izumisano, Osaka
  - Minoh City Hospital, Mino, Osaka
  - Kitano Hospital, Osaka, Osaka
  - Osaka City Juso Hospital, Osaka, Osaka
  - Osaka City General Hospital, Osaka, Osaka
  - Otemae Hospital, Osaka, Osaka
  - Osaka Police Hospital, Osaka, Osaka
  - Higashi Sumiyoshi Morimoto Hospital, Osaka, Osaka
  - Nissay Hospital, Osaka, Osaka
  - Osaka Kosei Nenkin Hospital, Osaka, Osaka
  - Osaka General Medical Center, Osaka, Osaka
  - Osaka Saiseikai Noe Hospital, Osaka, Osaka
  - Minamiosaka Hospital, Osaka, Osaka
  - Osaka Rosai Hospital, Sakai-shi, Osaka
  - Suita Municipal Hospital, Suita-shi, Osaka
  - Osaka Medical College, Takatsuki, Osaka
  - Saiseikai Tondabayashi Hospital, Tondabayashi, Osaka
  - Fukaya Red Cross Hospital, Fukaya, Saitama
  - Hasuda Hospital, Hasuda, Saitama
  - Saitama Medical School Hospital, Kawagoe-shi, Saitama
  - Saitama Social Insurance Hospital, Saitama, Saitama
  - National Defense Medical College, Tokorozawa, Saitama
  - Nagahama City Hospital, Nagahama, Shiga
  - Otsu Municipal Hospital, Ōtsu, Shiga
  - Shimane Prefectural Central Hospital, Izumo-shi, Shimane
  - Fujieda Municipal General Hospital, Fujieda, Shizuoka
  - Hamamatsu University School of Medicine, Hamamatsu, Shizuoka
  - Shizuoka City Hospital, Shizuoka, Shizuoka
  - Shizuoka Municipal Shimizu Hospital, Shizuoka, Shizuoka
  - Yaizu Municipal Hospital, Yaizu, Shizuoka
  - Jichi Medical School, Shimotsuke-shi, Tochigi
  - Tochigi Cancer Center, Utsunomiya, Tochigi
  - Anan Kyoei Hospital, Anan, Tokushima
  - St. Luke's International Hospital, Chuo-ku, Tokyo
  - Tokyo Metropolitan Fuchu Hospital, Fuchū, Tokyo
  - Shouwa General Hospital, Kodaira, Tokyo
  - Daisan Hospital, Komae, Tokyo
  - Kyorin University School of Medicine - Mitaka Campus, Mitaka, Tokyo
  - Social Insurance Chuo General Hospital, Shinjuku-ku, Tokyo
  - Tokyo Women's Medical University, Shinjyuku-ku, Tokyo
  - Mita Hospital at the International University of Health and Welfare, Tokyo, Tokyo
  - Tokyo Medical and Dental University, Tokyo, Tokyo
  - Nippon Medical School, Tokyo, Tokyo
  - Toho University School of Medicine, Tokyo, Tokyo
  - Japanese Red Cross Medical Center, Tokyo, Tokyo
  - International Medical Center of Japan, Tokyo, Tokyo
  - Teikyo University School of Medicine, Tokyo, Tokyo
  - Itabashi Chuo Medical Center, Tokyo, Tokyo
  - Takasago Kyoritsu Hospital, Tokyo, Tokyo
  - Tottori University - Faculty of Medicine, Yonago, Tottori
  - Koseiren Takaoka Hospital, Takaoka-shi, Toyama
  - Social Insurance Kinan Hospital, Tanabe, Wakayama
  - Yamagata Prefectural Central Hospital, Yamagata, Yamagata
  - Yamagata University Hospital, Yamagata, Yamagata
  - National Hospital Organization - Kanmon Medical Center, Shimonoseki, Yamaguchi
  - Shimonoseki Kosei Hospital, Shimonoseki, Yamaguchi
  - Yamaguchi University Graduate School of Medicine, Ube, Yamaguchi
  - University of Yamanashi Faculty of Medicine, Chu-o-shi, Yamanashi
  - Osaka Red Cross Hospital, Osaka